CLINICAL TRIAL: NCT06295172
Title: A Randomized, Evaluator-blind, Matched Pairs, Prospective, Non Inferiority, Confirmatory Study to Compare the Safety and Efficacy Between Lafullen15 and Lafullen in the Correction of Nasolabial Folds
Brief Title: A Study Comparing Lafullen15 and Lafullen for Temporary Nasolabial Fold Improvement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LF15_NLF_301
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-02

CONDITIONS: Nasolabial Folds

STUDY DESIGN:
Intervention Model Description: A Randomized, Evaluator-blind, Matched pairs, Prospective, Non inferiority, Confirmatory Study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lafullen15 (Experimental): PCL filler
  Interventions: Device: Lafullen15
- Lafullen (Active Comparator): PCL filler
  Interventions: Device: Lafullen

INTERVENTIONS:
Device: Lafullen15 — Apply a maximum of 1.0 ml for each side of the nasolabial fold using both the test device (Lafullen15) and the control device (Lafullen).
  Arms: Lafullen15
Device: Lafullen — Apply a maximum of 1.0 ml for each side of the nasolabial fold using both the test device (Lafullen15) and the control device (Lafullen).
  Arms: Lafullen

SUMMARY:
The objective of this clinical trial is to verify the safety and efficacy of Lafullen15 in the temporary improvement of nasolabial Folds

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who desire an improvement in the appearance of the nasolabial fold on both sides of the face and who have a score of 3 or 4 on the Wrinkle Severity Rating Scale (WSRS)
2. Individuals who have consented to abstain from any other dermatological procedures or treatments, including treatments for wrinkle reduction in the facial area, during the duration of this study

Exclusion Criteria:

1. Administered an anticoagulant (with the exception of low dosage aspirin (100mg, up to 300mg/day)) within 2 weeks of the date of the screening
2. Administered Vitamin E or non-steroidal anti-inflammatory drugs or Collagen within 1 week of the date of the screening, or who require these during the period of the study
3. History of bleeding disorder in past or present
4. Received deep-peeling, skin regeneration, plastic surgery (including botulinum toxin injection), wrinkle improvement or acne scar treatment in the facial area within 24 weeks of the date of the screening
5. Administered an hyaluronic acid filler within 24 weeks of the date of the screening

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2024-05-27 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in WSRS at 12 months after the last application of the clinical trial medical device compared to the baseline evaluated by an independent evaluator | 12months
  The Wrinkle Severity Rating Scale is a 5-point scale with 1 = Absent; 2 = Mild; 3 = Moderate; 4 = Severe and 5 = Extreme. 1 is the best outcome while 5 is the worst outcome. The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jongho KIM, M.D.,Ph.D., Principal Investigator — Seoul National University Bundang Hospital